CLINICAL TRIAL: NCT05314439
Title: A Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of Monthly Subcutaneous Administration of ION904 in Patients With Uncontrolled Hypertension
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of Monthly Subcutaneous Administration of ION904 in Participants With Uncontrolled Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ION904-CS2; 2022-000140-30 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ION904 (Experimental): Up to 4 monthly doses of ION904 will be administered by subcutaneous (SC) injection.
  Interventions: Drug: ION904
- Placebo (Placebo Comparator): Up to 4 monthly doses of placebo will be administered by SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ION904 — ION904 will be administered by SC injection.
  Arms: ION904
Drug: Placebo — Placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of ION904 on plasma angiotensinogen (AGT) in participants with uncontrolled hypertension.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, double-blind, randomized, placebo-controlled study. It will include up to approximately 48 participants with mild to moderate hypertension who have uncontrolled blood pressure (˃ 130 - ≤ 170 millimeters of mercury [mmHg] systolic) and have been on one or more anti-hypertensive medications for at least one month. Following an up to 4-week screening period, eligible participants will receive multiple doses of ION904 during a 13-week treatment period, followed by a 13-week post-treatment follow-up period.

ELIGIBILITY:
General Inclusion Criteria:

1. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential (WOCBP), she uses a highly effective contraceptive method. Aged 18 - 75 inclusive and weighing ≥ 50 kilograms (kg) at the time of informed consent
2. Body mass index (BMI) ≤ 45.0 kilograms per square meter (kg/m^2) at screening
3. History of uncontrolled hypertension (HTN) on one or more antihypertensive medications without changes in antihypertensive regimen within 4 weeks of screening and will be required to maintain this regimen throughout the Treatment Period

General Exclusion Criteria:

1. History of secondary HTN including, but not limited to any of the following: renovascular HTN (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug induced HTN
2. Unstable/underlying known cardiovascular disease defined as:

   * Any history of congestive heart failure (New York Heart Association [NYHA] Class III-IV)
   * Any history of previous myocardial infarction, coronary revascularization, unstable or stable angina pectoris ˂ 6 months prior to screening
   * Any hemodynamically unstable atrial or ventricular arrhythmias
   * Significant uncorrected valvular heart disease
   * Any history of stroke or transient ischemic attack < 6 months prior to screening
3. A cardiac valve repair, cardiac device implantation, and/or a hospitalization for heart failure within 3 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Plasma Angiotensinogen (AGT) | Baseline up to approximately 15 weeks

SECONDARY OUTCOMES:
Change from Baseline in Seated Automated Office Systolic Blood Pressure (SBP) | Baseline up to approximately 15 weeks
Change from Baseline in Seated Automated Office Diastolic Blood Pressure (DBP) | Baseline up to approximately 15 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Altasciences - Los Angeles, Cypress, California
  - National Research Institute, Los Angeles, California
  - Clinical Trials Research, Sacramento, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Altasciences, Overland Park, Kansas
  - NY Scientific, Brooklyn, New York
  - Juno Research, LLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No